CLINICAL TRIAL: NCT00202670
Title: Diagnosis of Coronary Artery Disease in High Risk Diabetic Patients :Comparison Between Stress Echocardiography and Stress Scintigraphy in the Detection of Silent Myocardial Ischemia
Brief Title: Diagnosis of Coronary Artery Disease in High Risk Diabetic Patients
Status: Terminated | Type: Observational
Why Stopped: Positive Predictive value not related to follow up duration.
Sponsor: Société Française de Cardiologie (Other)
Responsible Party: Société Françaisede Cardiologie
Other Study IDs: 2003-04
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2010-10-20 (Estimated); Status verified 2004-01

CONDITIONS: Diabetes Mellitus
Keywords: coronary artery disease; stress myocardial scintigraphy; stress echocardiography
MeSH Terms: conditions — Diabetes Mellitus; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1: SPECT
- 2: dobutamine echocardiography

SUMMARY:
The aim of this study is to determine in high risk diabetics if the positive predictive value of stress echocardiography is superior to the positive predictive value of stress scintigraphy in the diagnosis of coronary stenosis > 50%.

DETAILED DESCRIPTION:
Comparison Between Stress Echocardiography and Stress Scintigraphy in the Detection of Silent Myocardial Ischemia

ELIGIBILITY:
Inclusion Criteria:

* type 2 diabetic patients in women> 60 yo or men > 55 yo, with high risk of coronary artery disease (EF < 40%, ECG abnormalities, renal failure , 2 others risk factors of atherosclerosis)

Exclusion Criteria:

* previous documented CAD acute coronary syndrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: high risk diabetic patients
Sampling Method: Probability Sample
Enrollment: 220 (Estimated)
Dates: Start 2004-01; Primary Completion 2010-05 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Claude Le Feuvre, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (2):
- France (2):
  - Pitie Salpetriere, Paris
  - Service de diabétologie - Pitié Salpêtrière, Paris

REFERENCES:
- [Derived] Jacqueminet S, Barthelemy O, Rouzet F, Isnard R, Halbron M, Bouzamondo A, Le Guludec D, Grimaldi A, Metzger JP, Le Feuvre C. A randomized study comparing isotope and echocardiography stress testing in the screening of silent myocardial ischaemia in type 2 diabetic patients. Diabetes Metab. 2010 Dec;36(6 Pt 1):463-9. doi: 10.1016/j.diabet.2010.06.005. Epub 2010 Sep 15. PMID 20832344